CLINICAL TRIAL: NCT07353268
Title: A Phase Ib/II Study Evaluating the Safety, Tolerability, and Efficacy of Epalolitovoreli Monoclonal Antibody (QL1706) and Fruquintinib Combined With Short-Course Radiotherapy (SCRT) Versus Standard Third-Line Therapy in Patients With Unresectable Liver-Metastatic pMMR/MSS Colorectal Cancer.
Brief Title: Phase Ib/II Study of QL1706 + Fruquintinib + SCRT vs. Standard Third-Line Therapy in Unresectable Liver-Metastatic pMMR/MSS Colorectal Cancer: Safety, Tolerability, and Efficacy.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tao Zhang (Other)
Responsible Party: Sponsor-Investigator, Tao Zhang, MD, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZLK20250622
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL1706 + Fruquintinib + Short-Course Ablative Radiotherapy (SCART) (Experimental): Patients will receive the PD-1/CTLA-4 bispecific antibody Epalolitovoreli Monoclonal Antibody (QL1706) at a dose of 5 mg/kg by intravenous infusion every 3 weeks (Q3W).
  Patients will concomitantly receive oral Fruquintinib once daily (QD). The dose will be determined in a Phase Ib dose-escalation phase exploring 3 mg and 4 mg QD levels, using a modified 3+3 design to establish the Recommended Phase II Dose (RP2D).
  Patients will undergo Short-Course Ablative Radiotherapy (SCART) to the liver metastasis/metastases. The prescribed dose is 15 Gy in 3 fractions to the Gross Tumor Volume (GTV) and 45-72 Gy in 3 fractions to the Subclinical Target Volume (STV).
  Treatment with QL1706 and Fruquintinib will continue until disease progression, unacceptable toxicity, or other protocol-specified discontinuation criteria.
  Interventions: Drug: QL1706 + Fruquintinib + Short-Course Ablative Radiotherapy (SCART)
- Standard Third-Line Therapy (Active Comparator): Patients will receive one of the following standard-of-care third-line therapies for metastatic colorectal cancer, selected by the investigator based on the patient's prior treatment history and comprehensive condition:
  Cetuximab with or without Irinotecan (for patients not previously treated with cetuximab).
  Regorafenib. Fruquintinib. Trifluridine/Tipiracil (TAS-102) with or without Bevacizumab.
  Interventions: Drug: Standard Third-Line Therapy

INTERVENTIONS:
Drug: QL1706 + Fruquintinib + Short-Course Ablative Radiotherapy (SCART) — Patients will receive the PD-1/CTLA-4 bispecific antibody Epalolitovoreli Monoclonal Antibody (QL1706) at a dose of 5 mg/kg by intravenous infusion every 3 weeks (Q3W).
  Patients will concomitantly receive oral Fruquintinib once daily (QD). The dose will be determined in a Phase Ib dose-escalation phase exploring 3 mg and 4 mg QD levels, using a modified 3+3 design to establish the Recommended Phase II Dose (RP2D).
  Patients will undergo Short-Course Ablative Radiotherapy (SCART) to the liver metastasis/metastases. The prescribed dose is 15 Gy in 3 fractions to the Gross Tumor Volume (GTV) and 45-72 Gy in 3 fractions to the Subclinical Target Volume (STV).
  Treatment with QL1706 and Fruquintinib will continue until disease progression, unacceptable toxicity, or other protocol-specified discontinuation criteria.
  Arms: QL1706 + Fruquintinib + Short-Course Ablative Radiotherapy (SCART)
Drug: Standard Third-Line Therapy — Patients will receive one of the following standard-of-care third-line therapies for metastatic colorectal cancer, selected by the investigator based on the patient's prior treatment history and comprehensive condition:
  Cetuximab with or without Irinotecan (for patients not previously treated with cetuximab).
  Regorafenib. Fruquintinib. Trifluridine/Tipiracil (TAS-102) with or without Bevacizumab.
  Arms: Standard Third-Line Therapy

SUMMARY:
This study is designed to evaluate the safety, tolerability, and efficacy of Epalolitovoreli Monoclonal Antibody (QL1706) combined with Fruquintinib and Short-Course Radiotherapy (SCRT), compared with standard third-line therapy, in the treatment of patients with unresectable liver-metastatic pMMR/MSS colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent, and ability to comply with the scheduled visits and related procedures as specified in the protocol.
2. Age ≥18 years and ≤75 years, male or female.
3. Histologically or cytologically confirmed metastatic colorectal cancer with unresectable liver metastasis(es) measuring ≥5 cm in the longest diameter.
4. Confirmed pMMR (proficient mismatch repair) or MSS (microsatellite stable) status by immunohistochemistry (IHC), next-generation sequencing (NGS), or PCR testing.
5. Disease progression after, intolerance to, lack of access to, or refusal of standard second-line therapy.
6. Baseline* hematologic tests (within 7 days prior to the first dose of study drug) meeting the following criteria:

   * Hemoglobin ≥90 g/L.
   * Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L.
   * Platelet count ≥100 × 10⁹/L.
   * Eosinophil count ≤1.5 × Upper Limit of Normal (ULN).
7. Baseline serum biochemical tests (within 7 days prior to the first dose) meeting the following criteria:

   * Total bilirubin ≤1.5 × ULN (if total bilirubin >1.5 × ULN but direct bilirubin ≤ ULN, enrollment is permitted).
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤3 × ULN.
   * Serum creatinine ≤1.5 × ULN or creatinine clearance (CCr) ≥45 mL/min (calculated using the Cockcroft-Gault formula with actual body weight).
   * Albumin ≥30 g/L.
8. Baseline coagulation tests (within 7 days prior to the first dose) meeting the following criteria:

   * International normalized ratio (INR) ≤1.5 × ULN (or ≤3 × ULN if on stable-dose anticoagulation therapy).
   * Partial thromboplastin time (PTT) [or activated partial thromboplastin time (aPTT)] ≤1.5 × ULN (or ≤3 × ULN if on stable-dose anticoagulation therapy).
9. Baseline urinalysis (within 7 days prior to the first dose) meeting the following criterion: Urine protein (UPRO) <2+ or 24-hour urine protein quantification <1 g.
10. At least one measurable lesion as defined by RECIST v1.1 criteria.
11. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
12. Life expectancy ≥3 months.
13. For female patients of childbearing potential or male patients with partners of childbearing potential, agreement to use effective contraception strictly throughout the treatment period and for 6 months thereafter.

Exclusion Criteria:

* 1. History of allergy to any study drug, including Epalolitovoreli Monoclonal Antibody and Fruquintinib.

  2. Pregnant or breastfeeding women, or women planning to become pregnant within 6 months before, during, or after the last dose of study drug.

  3. Known history of active seizures, active central nervous system metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal metastases; newly diagnosed brain or leptomeningeal metastases.

  4. Cardiovascular or cerebrovascular diseases with significant clinical implications, including:
  * Ventricular arrhythmias or other uncontrolled arrhythmias requiring medical intervention (e.g., antiarrhythmic medication).
  * Severe conduction disorders (e.g., third-degree atrioventricular block).
  * Heart rate-corrected QT interval (QTc, calculated using Fridericia's formula) ≥480 ms.
  * Uncontrolled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg), history of hypertensive crisis or hypertensive encephalopathy.
  * History of myocarditis.
  * Current congestive heart failure requiring treatment.
  * New York Heart Association (NYHA) Class III or IV cardiovascular disease.
  * Acute coronary syndrome (including myocardial infarction and unstable angina), coronary angioplasty, or stenting within 6 months prior to the first dose.
  * Cerebrovascular accident or transient ischemic attack within 6 months prior to the first dose.
  * Interstitial lung disease, pulmonary fibrosis, pneumoconiosis, drug-related pneumonia, radiation pneumonitis requiring steroid or other treatment, severe pulmonary dysfunction, or history of other forms of restrictive lung disease.

    5. History of allergic constitution, asthma, or atopic dermatitis. 6. Patients with massive pleural effusion or massive ascites. 7. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary insufficiency) is not considered systemic treatment.

    8. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

    9. Known or suspected hypersensitivity to the study drugs or any of their excipients.

    10. History of significant toxicity related to immune checkpoint inhibitors or Fruquintinib-class drugs that led to permanent discontinuation of the treatment.

    11. Residual toxicity > Grade 1 from any prior anti-tumor therapy (except for persistent Grade 2 alopecia, peripheral neuropathy, decreased hemoglobin, and hypomagnesemia).

    12. Active uncontrolled bleeding, known bleeding tendency, severely unhealed wounds, ulcers, or fractures; such as esophageal or gastric varices requiring immediate intervention (e.g., ligation or sclerotherapy); or evidence of portal hypertension deemed by the investigator to confer a high risk of bleeding.

    13. Patients with risk of bowel obstruction (except surgically cured or completely resolved obstruction) or gastrointestinal perforation within 28 days prior to the first dose in this study (including, but not limited to, acute diverticulitis, intra-abdominal abscess, abdominal cancer, history of gastrointestinal perforation and/or fistula within 6 months prior to screening).

    14. Patients with current or recent (within 6 months) significant gastrointestinal disease or conditions, including:

    a) History of clinically significant gastrointestinal bleeding. b) Active peptic ulcer. c) Diarrhea ≥ Grade 2 within 2 weeks prior to the first dose. 15. Patients with uncontrolled tumor-related pain or symptomatic hypercalcemia. 16. Known positive HIV test, active Hepatitis B, Hepatitis C (HCV), tuberculosis, or history of such infections. Exceptions are as follows:
  * Patients who are HBsAg positive or HBcAb positive must have HBV DNA ≤2.5 × 10³ copies/mL or ≤500 IU/mL or below the limit of detection to be eligible.
  * Patients with positive HCV serology are eligible if HCV RNA is negative or below the limit of detection.
  * Patients who have received HCV treatment and have undetectable viral loads are eligible.

    17. Severe/active/uncontrolled infection requiring systemic intravenous antibiotic therapy, or unexplained fever (>38°C) within 2 weeks prior to the first dose.

    18. Diagnosis of another malignancy within 5 years prior to the first dose, except for radically treated basal cell carcinoma, squamous cell carcinoma of the skin, radically resected carcinoma in situ, radically treated localized prostate cancer, papillary thyroid carcinoma, etc.

    19. Prohibited medications and other treatments (patients must not receive any of the following):
  * Any chemotherapy or small molecule targeted therapy within 2 weeks or 5 half-lives (whichever is shorter) prior to the first dose, without delayed toxicity.
  * Any monoclonal antibody therapy within 4 weeks prior to the first dose.
  * Participation in any interventional clinical trial involving medical devices or other therapies within 2 weeks prior to the first dose.
  * Palliative radiotherapy within 2 weeks prior to the first dose.
  * Live vaccines for infectious disease prevention within 4 weeks prior to the first dose.
  * Immunosuppressive or systemic corticosteroid therapy (>10 mg/day prednisone equivalent) within 2 weeks prior to the first dose.
  * For patients on anticoagulant therapy, coagulation parameters are not stably controlled within the target range, or there is unstable thrombosis, pulmonary embolism events, or clinically significant bleeding events within the past 6 months.
  * Any major surgery within 4 weeks prior to the first dose. 20. Any disease, treatment, laboratory abnormality, history of substance abuse, or current evidence that, in the investigator's judgment, may compromise the patient's safety, interfere with obtaining informed consent, affect patient compliance, or impact the safety evaluation of the study drug.

    21. Patients deemed unsuitable for participation in this study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival（PFS） | an expected average of 6 months
  Progression-free survival (PFS) is defined as the time from the initiation of study treatment to the first occurrence of disease progression or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival | an expected average of 5 years
  The time from the date of randomization to the death caused by any cause
dverse events (AEs) were graded according to the NCI CTCAE version 5·0 | an expected average of 1.5 years
  Adverse events and surgical safety

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided